CLINICAL TRIAL: NCT07361172
Title: Ready-made vs. Custom-made Carriere Motion Appliance: A Randomized Clinical Trial
Brief Title: Ready-made vs. Custom-made Carriere Motion Appliance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0101025OR
Record Dates: First submitted 2025-08-10; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Class II Malocclusion
Keywords: Class II malocclusion; Carriere motion appliance; Distalization
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-made CMA (Experimental): Custom-made CMA from brackets, buccal tubes, stiff wire, and NiTi coil springs
  Interventions: Device: Custom-made Carriere motion appliance
- Ready-made CMA (Active Comparator)
  Interventions: Device: Ready-made Carriere motion appliance

INTERVENTIONS:
Device: Custom-made Carriere motion appliance — custom-made CMA from brackets, buccal tubes, stiff wire, and NiTi coil springs to treat class II malocclusion by molar distalization.
  Arms: Custom-made CMA
Device: Ready-made Carriere motion appliance — Ready-made Carriere motion appliance to treat class II malocclusion by molar distalization.
  Arms: Ready-made CMA

SUMMARY:
The aim of this study is to evaluate the effect of custom-made CMA vs. the ready-made CMA.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of custom-made CMA from brackets, buccal tubes, stiff wire, and NiTi coil springs and compare it with the ready-made CMA.

ELIGIBILITY:
Inclusion Criteria:

* Patients age (12-15) years.
* Full permanent dentition.
* Class II malocclusion with at least an end-on Class II molar relationship bilaterally.

Exclusion Criteria:

* Systemic conditions that may interfere with the treatment.
* Bad habits that might jeopardize the appliance.
* Transverse discrepancy.
* Previous orthodontic treatment.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Treatment duration | up to 6 months from the start of treatment until the date of first documented progression
  in about 6 months from the start of treatment till reaching class I molar relation
Skeletal and dental changes | up to 6 months from the start of treatment until the date of first documented progression
  angular and linear cephalometric measurements

SECONDARY OUTCOMES:
Soft tissue changes | up to 6 months from the start of treatment until the date of first documented progression
  angular and linear cephalometric measurements
Patient satisfaction | up to 6 months from the start of treatment until the date of first documented progression
  patient questionnaire about oral health related quality of life: their satisfaction and discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Adakhlia, Egypt